CLINICAL TRIAL: NCT01233570
Title: Topical Tacrolimus 0.1% Ointment for Treatment of Cutaneous Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Dr AD Ormerod, University of Aberdeen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33000332
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Crohn Disease
Keywords: Cutaneous Crohns Disease; Topical Tacrolimus; Protopic; Metastatic Crohns Disease; Pyoderma Gangrenosum; Granulomatous chelitis; Oral crohns disease; Perianal crohns disease
MeSH Terms: conditions — Crohn Disease; Pyoderma Gangrenosum | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topical tacrolimus (Experimental): Once daily topical application
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Once daily application for 12 weeks followed by 4 weeks observation. Optional 36 week open label extension
  Other Names: Protopic 0.1%; FK506

SUMMARY:
An assessment of the efficacy of topical tacrolimus in the treatment of cutaneous crohns disease

ELIGIBILITY:
Inclusion Criteria:

* willingness and capability to follow the study procedure
* confirmed diagnosis of Crohn's Disease of at least 3 months duration confirmed by radiography, endoscopy or pathological examination
* required to have a skin manifestation of Crohn's disease
* required to give written informed consent
* both male and female subjects with reproductive potential required to be on an acceptable form of birth control for the duration of the study
* long-standing, concomitant immunosuppressive therapy was allowed if the dose was stable and not controlling the skin problem

Exclusion Criteria:

* known sensitivity to tacrolimus
* change in aminosalicylate dosage in the four weeks prior to screening
* on oral steroids at over 40mg per day
* been commenced on methotrexate, azathoprine or ciclosporin within the last two months
* commenced on a a TNF-alpha monoclonal antibody within the three months prior to screening
* patients having had a stoma fashioned less than three months before enrolment
* patients with an immunocompromising disease
* patients with a diagnosis of malignancy within the last five years
* patients with any other condition, past or present treatment thought by the investigator to render the subject ineligible for the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)

PRIMARY OUTCOMES:
Assessment of standardised digital photography by three independent assessors following the Physicians' Global Severity Scale before and after treatment | At 12 weeks of treatment, optionally extended to 52 weeks

SECONDARY OUTCOMES:
Global Self Assessment | 12 weeks, optionally extended to 52 weeks
Perineal Disease Activity Index | 12 weeks, optionally extended to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Ormerod, MBChB, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen Royal Infirmary, Aberdeen, Grampian, United Kingdom